CLINICAL TRIAL: NCT02903615
Title: The Optimal Diet for Optimising Health in Type 1 Diabetes
Brief Title: Optimising Health in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Garvan Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Professor Katherine Samaras, Professor, Garvan Institute of Medical Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/053
Record Dates: First submitted 2016-06-05; First posted 2016-09-16 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus
Keywords: glucose; inflammation
MeSH Terms: conditions — Diabetes Mellitus; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Novel type 1 diet (Experimental): Experimental diet to be examined: altered macronutrient composition: lower carbohydrate, Mediterranean-style, prebiotic fibre focus.
  Interventions: Other: Novel diet
- Standard therapy (Placebo Comparator): Standard dietary therapy, as promulgated by Australian standards
  Interventions: Other: Standard diet

INTERVENTIONS:
Other: Novel diet — Novel diet to optimise glucose levels and minimise systemic inflammation: altered macronutrient composition: lower carbohydrate, Mediterranean-style, prebiotic fibre focus.
  Arms: Novel type 1 diet
Other: Standard diet — Standard diabetes diet recommendations
  Arms: Standard therapy

SUMMARY:
Type 1 diabetes is an autoimmune condition where circulating immune cells destroy the beta-cells in the pancreas that make insulin, resulting in a degree of insulin deficiency, whereby blood glucose levels rise and diabetes develops. When there is severe insulin deficiency, life-threatening ketoacidosis can develop. Treatment is lifelong insulin replacement therapy; dietary intervention is a also cornerstone of glucose management.

The Optimise Diet is a multi-pronged diet based on "best health" principles: to minimise blood glucose rises after eating, reduce the immune cells involved in destruction of the insulin-secreting beta-cells, and improve the gut microbiome and systemic inflammation. In this study, its effects will be compared to the Standard Diabetes Diet that is currently recommended in Australia and internationally.

DETAILED DESCRIPTION:
The rationale for this study is to determine whether a diet based on recent scientific advances in diet-induced inflammation, will improve diabetes care in people with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes

Exclusion Criteria:

* Women lactating, pregnant or of childbearing potential who are not willing to avoid becoming pregnant during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Glucose control | 3 months
  HbA1c

SECONDARY OUTCOMES:
Inflammation | 3 months
  Circulating immune cells numbers
Gut microbiome | 3 months
  Gut flora subtypes
C-peptide | 3 months
  Urinary excretion
postprandial glucose excursion | 3 months
  postprandial glucose excursion
Follow-up of glycemic control and insulin secretion | 12 and 24 months
  HbA1c, urinary C-peptide

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Samaras, MD PhD FRACP, Principal Investigator — Garvan Institute of Medical Research
Locations (2):
- Australia (2):
  - professor Katherine Samaras, Sydney, New South Wales
  - Garvan Institute to Medical Research, Sydney

IPD SHARING:
Plan to Share IPD: Undecided